CLINICAL TRIAL: NCT00518193
Title: Phase II Study , Association of Cisplatine Topotecan and Cetuximab in Patients Whith Late or in Progress Epithelial Cancer of the Cervix
Acronym: ERBUS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: high rate of medullar aplasia with infectious troubles.
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Frédéric MARMION, ARCAGY-GINECO
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERBUS
Record Dates: First submitted 2007-08-14; First posted 2007-08-20 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ERBITUX — 400 mg/m² 2h injection at week 1, then 250 mg/m² in one hour injection the following weeks

SUMMARY:
The efficacy of chimiotherapy in cervix epithelial cancer is low even with the association cisplatine - topotecan .

News thérapeutics are needed in the goal of increase the survival and quality of life in patients with cervix cancer.

Cetuximab has shown the potentialisation on the efficacy of cisplatine and irinotecan.

Cisplatine and topotecan have shown an efficacy in cervix cancer. Cetuximab is well tolerate. Many clinical trials shown the faisability of the association of cetuximab and cisplatine in cancer.

Many clinical trials have shown the faisability of association of cetuximab and irinotecan in colorectals metastatiques cancers .

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old.
* Epidermoïde carcinoma or adenocarcinoma of the cervix, hystologic proved
* Patientes in a late stage or with progresive desease.
* One mesurable lesion in irradiated zone.
* Patient who have already treated radio-chimiothérapy with platine should have a 6 month free interval.
* Index status of ECOG (" Eastern Cooperative Oncology Group ")less than 2.
* Good biologicals and hematologicals fonctions:
* Neutrophiles noless than 1,5.109/L.
* Platelets nolss than 100.109/L.
* Total bilirubin no more than 1,5 time the normal superior range.
* Transaminases no mote than 3 x Time NSR
* Creatinine clairance Cockroft) more than 50 mL/min .
* Inform consent signed.

Exclusion Criteria:

* Previous cytotoxic traitement exept radio-chaemiotherapy of the pelvis cerebrals metastasis.
* Other cancer in the last 5 years exept treated BCC.
* Dermatologic desease.
* Crohn desease or Hemorragic rectal-Colitis.
* Neuropathy.
* Psychologic disorder.
* Social troubles.
* Pregnant women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-04; Primary Completion 2007-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
responses rate regarding the RECIST criteria. | up to progression

SECONDARY OUTCOMES:
Quality of life, free interval, safety. | up to progression

CONTACTS AND LOCATIONS:
Overall Officials: Pr KURTZ Jean Emmanuel, Principal Investigator — STRASBOURG
Locations (4):
- France (4):
  - CRLC Val d'Aurelle, Montpellier
  - Hôpital HOTEL DIEU, Paris
  - Oncologie, Hôtel-Dieu, 1 place du parvis Notre-Dame, Paris
  - Centre Claudius Régaud, Toulouse

REFERENCES:
- See also: Related Info — http://www.arcagy.org